CLINICAL TRIAL: NCT00828893
Title: Interest of the Use of a Navigation Guidance Gestures Carried Out Under CT
Brief Title: Navigation Guidance Gestures Carried Out Under CT
Acronym: CT-Nav
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AdministrateurCIC (Other)
Responsible Party: Sponsor-Investigator, AdministrateurCIC, principal investigator, University Hospital, Grenoble
Organization: University Hospital, Grenoble (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DCIC 08 01; IMACTIS company
Record Dates: First submitted 2009-01-23; First posted 2009-01-26 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Drainage; Biopsy; Punction
Keywords: drain under scanner

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: navigation station — navigation station for gestures (carried out under CT) guidance

SUMMARY:
The purpose of this study is to assess the contribution of navigation systems recently developed to guide the punction needle.

ELIGIBILITY:
Inclusion Criteria:

* more or equal than 18 years old
* patient affiliated to social security or similarly regime
* patient sent to hospital for drain under CT

Exclusion Criteria:

* Pregnant women and lactating mothers
* Ward of court or under guardianship
* Adult unable to express their consent
* Person deprived of freedom by judicial or administrative decision
* Person hospitalized without their consent
* Person under legal protection
* Person participating in another clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Maximum distance between the planned trajectory and trajectory achieved, defined for the needle of local anesthesia. | 2 hours

SECONDARY OUTCOMES:
Maximum distance between the planned trajectory and trajectory achieved by the needle puncture. | 2 hours
Duration of intervention | 3 hours
Dose irradiation and number of control scanners made | 3 hours
overall satisfaction Score | 3 hours
Success or failure of the final gesture made | 3 hours
Number of attempts | 3 hours
number of complications (per-operative, post-surgery) | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- UniversityHospitalGrenoble, Grenoble, France

REFERENCES:
- [Derived] Robert AL, Chagnon G, Bricault I, Cinquin P, Moreau-Gaudry A. A generic three-dimensional static force distribution basis for a medical needle inserted into soft tissue. J Mech Behav Biomed Mater. 2013 Dec;28:156-70. doi: 10.1016/j.jmbbm.2013.07.023. Epub 2013 Aug 9. PMID 23988636